CLINICAL TRIAL: NCT02252107
Title: 10-day Decitabine, Fludarabine and 2 Gray TBI as Conditioning Strategy for Poor and Very Poor Risk AML in CR1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLMA34
Record Dates: First submitted 2014-09-19; First posted 2014-09-29 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Decitabine; Hematopoietic stem cell transplantation (HSCT); Conditioning; AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine (Experimental): Single arm study: the addition of 10 days (20 mg/m2) decitabine to the conditioning regimen prior to allogeneic hematopoietic transplantation.
  Interventions: Drug: decitabine

INTERVENTIONS:
Drug: decitabine — Single arm study: the addition of 10 days (20 mg/m2) decitabine to the conditioning regimen prior to allogeneic hematopoietic transplantation.
  Other Names: Dacogen

SUMMARY:
This study examines whether the addition of decitabine to the standard Flu/TBI conditioning regimen prior to allogeneic stem cell transplantation in poor and very poor risk AML patients, reduces the risk of recurrence of the disease. Because decitabine has hardly any side effects, it will likely have little impact on the occurrence of Graft Versus Host Disease. The investigators are looking for a pre-treatment for transplantation which reduces the chance of recurrence of the disease without involving severe damage to normal tissues.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a heterogeneous group of malignant hematological diseases with different molecular genetic abnormalities. These are important in predicting response to treatment. Recently, an analysis of 424 AML patients treated in various HOVON protocols showed a 5 year overall survival for patients in good, intermediate, poor and very poor risk groups of 65%, 51%, 25% and 7% respectively (HOVON 102 protocol). This shows that especially for patients in the (very) poor risk group, the outcome is very disappointing, despite the current treatment strategies. For patients with intermediate, poor and very poor risk cytogenetics postconsolidation treatment with an allogeneic hematopoietic cell transplantation (allo HCT) is standard practice after myeloablative (MAB HCT) or non-myeloablative (NMA HCT) conditioning.

Unfortunately, mortality after MAB conditioning is still considerable, mainly due to therapy related mortality, graft-versus-host disease, infections, or relapse. Currently, the NMA conditioning is used more frequently, which is far less toxic. Nonmyeloablative regimens have relied on the immunological anti-leukemia effect (graft-versus-leukemia), to prevent relapsing disease. This anti-leukemia effect, however, needs time to develop, which makes it necessary to be in control over the disease pre-transplantation as much as possible. This extends the time the immune system of the donor has to develop an adequate anti-leukemia effect, which is especially important in the (very) poor risk group patients since they have the highest chance of relapse.

Epigenetic alterations are increasingly recognised for their roles in oncogenesis. These alterations can for example 'silence'genes by hypermethylation. These alterations are potentially reversible.

The hypomethylating agent decitabine is one of the therapeutic approaches which can reactivate silenced genes by its interaction on the epigenetics. A phase II study (Blum, Proc Natl Acad Sci 2010) with 53 AML patients who received 10 days decitabine, showed a complete remission rate (CR) in 47% of patients. This percentage corresponds to the CR of intensive chemotherapy in elderly AML patients. The median survival was 55 weeks. Furthermore, this study showed that decitabine was well tolerated.

Earlier studies have shown that patients whose disease was controlled with hypomethylating agents pre-transplantation had comparable survival compared with patients whose disease was controlled with intensive chemotherapy(Damaj, Journal of Clinical Oncology, 2012).

In the current study the AML is already in remission after intensive chemotherapy. In an attempt to design a conditioning strategy with very low toxicity but considerable myelosuppressive activity, the investigators will combine the non-myeloablative (NMA) fludarabine and low-dose TBI (2 Gray) with a 10-day schedule of decitabine (Dec-Flu-TBI). Theoretically, it is very attractive to add a drug like decitabine (in a 10-day schedule) that exerts a strong antileukemic effect, without additional extra-medullary toxicity, to the standard Flu-TBI NMA conditioning regimen. The hypothesis is that in this way the investigators can extent the time the immune system of the donor needs to create an adequate graft-versus-leukemia effect, at the cost of low toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for allogeneic HCT, independent of age
* Adult patients of any age with a cytopathologically confirmed diagnosis according to WHO classification of newly diagnosed AML (not APL = AML-M3), de novo AML or secondary AML
* in first complete remission (CR1)
* Poor risk or very poor risk subgroups
* WHO performance status ≤ 2
* Written informed consent

Exclusion Criteria:

* Patient not in CR1
* Patients who have senile dementia, mental impairment of any other psychiatric disorder that prohibits the patient from understanding and giving informed consent
* Active serious infections like HIV, hepatitis B virus (HBV) and hepatitis C virus (HCV)
* Patient is unwilling to use contraceptive techniques during and for 12 months following treatment
* Female patient who is pregnant or breastfeeding
* Active and uncontrolled infections

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Relapse at 1-year after the transplantation procedure | At 1-year after the transplantation procedure
  All patients included in this study are in complete morphologic remission. Relapse at 1-year is defined as the % of patients who have relapsed within the first year after transplantation. For the computation of the incidence of relapse at 1-year, death in CR will be considered as a competing risk.

SECONDARY OUTCOMES:
Relapse within the first 100 days after the transplantation procedure | 100 days after the transplantation procedure
  All patients included in this study are in complete morphologic remission. Relapse within the first 100 days after the transplantation procedure is defined as the % of patients who have relapsed within the first100 days after the transplantation procedure. For the computation of the incidence of relapse within 100 days after the transplantation procedure, death in CR will be considered as a competing risk.
Treatment related mortality (TRM) within the first 100 days after the transplantation procedure | 100 days after the transplantation procedure
  Treatment related mortality (TRM) within the first 100 days after the transplantation procedure is defined as the % of patients deceased related to the treatment/whereby death is related to the treatment, within the first 100 days after the transplantation procedure.
Treatment related mortality (TRM) at 1-year after the transplantation procedure | At 1-year after the transplantation procedure
  Treatment related mortality (TRM) at 1-year after the transplantation procedure is defined as the % of patients deceased related to the treatment/whereby death is related to the treatment, within the first year after the transplantation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Gerwin Huls, MD. PhD., Principal Investigator — Radboud University Medical Center
Locations (3):
- University of Liège, Liège, Belgium
- Netherlands (2):
  - University Medical Center Groningen (UMCG), Groningen
  - Radboud university medical center, Nijmegen

REFERENCES:
- [Derived] Cruijsen M, Hilberink JR, van der Velden WJFM, Jansen JH, Bar B, Schaap NPM, de Haan A, Mulder AB, de Groot MR, Baron F, Vellenga E, Blijlevens NNM, Huls G. Low relapse risk in poor risk AML after conditioning with 10-day decitabine, fludarabine and 2 Gray TBI prior to allogeneic hematopoietic cell transplantation. Bone Marrow Transplant. 2021 Aug;56(8):1964-1970. doi: 10.1038/s41409-021-01272-3. Epub 2021 Apr 6. PMID 33824442